CLINICAL TRIAL: NCT03015480
Title: Facilitating Improvements in Kidney Health Using a Smartphone App Counseling Program in Patients With Diabetes
Acronym: FitKidney
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geisinger Clinic (Other)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2016-0382
Record Dates: First submitted 2017-01-04; First posted 2017-01-10 (Estimated); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Chronic Kidney Disease; Diabetes Mellitus; Albuminuria
Keywords: Mobile Application; Chronic Kidney Disease; Diabetes Mellitus; Albuminuria; Diet
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetes Mellitus; Albuminuria

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Remote counseling (Experimental): This group of people will be asked to track dietary information on MyFitnessPal and receive remote dietary counseling with a dietitian.
  Interventions: Behavioral: Remote counseling

INTERVENTIONS:
Behavioral: Remote counseling — For an 8 week period, patients will be asked to enter dietary information into the MyFitnessPal mobile application or website. Dietitians will access this information and provide personalized motivational interview phone calls on a weekly basis. After the initial 8 weeks, patients will receive a dietitian follow-up phone call around 5 and 11 months later.

SUMMARY:
This pilot study tests the feasibility of dietary app-supported tele-counseling in the treatment of patients with stage 1-3a chronic kidney disease (CKD) and diabetes.

DETAILED DESCRIPTION:
Patients with diabetes and stage 1-3a CKD receive instructions on downloading and using MyFitnessPal on their smartphone or computer to log meal data daily, weekly website educational materials, and weekly telephone visits with a dietician for 8 weeks. Patients receive a follow-up phone call from the dietitian and 5 and 11 months for further support and counseling, and are also invited to attend a local dietitian-led grocery tour. This pilot study examines the feasibility of dietary app-supported tele-counseling in the treatment of patients with stage 1-3a chronic kidney disease (CKD) and diabetes.

Main outcomes include sodium intake assessed by 24 hour urine collection as well as other dietary measures related to kidney disease (sodium/potassium ratio, Healthy Eating Index score, 24-hour urine phosphorus, estimated net endogenous acid production) and health measures (24-hour ambulatory blood pressure, weight, albumin/creatinine ratio)

ELIGIBILITY:
Inclusion Criteria:

* Age > 21 years
* Diabetes diagnosis (Type I or Type II)
* Last urine albumin/creatinine ratio (ACR) within the past two years > 30 mg/g
* Last outpatient estimated glomerular filtration rate (eGFR) within the past year > 45 ml/min/1.73m2
* Last outpatient systolic blood pressure (SBP) within the past year < 160 mmHg
* Last outpatient diastolic blood pressure (DBP) within the past year <100 mmHg
* Preceding eGFR decline rate less than -2 ml/min/1.73m2/y
* At least 2 outpatient eGFR measurements in electronic health record, separated by at least 2 years
* Agreeable to change diet (decrease sodium and red/processed meat intake, increase fruit and vegetable intake)
* Access to smartphone or computer

Exclusion Criteria:

* Inability to understand English
* Myocardial infarction, stroke, or atherosclerotic cardiovascular disease procedure within 6 months.
* Current treatment for malignancy
* Planned bariatric surgery
* Pregnancy or planning to become pregnant within next 2 years
* Self-reported average consumption of > 14 alcoholic beverages per week
* Psychiatric hospitalization in past year
* Unstable angina
* Urine ACR > 2500 mg/g
* Last potassium > 5.0 mg/dL
* Hypoglycemia episode in past 1 month (glucose < 70 mg/dL)
* Principal investigator discretion (i.e. concerns about safety, compliance)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-02-13 (Actual); Primary Completion 2018-11-25 (Actual); Study Completion 2018-11-25 (Actual)

PRIMARY OUTCOMES:
Change in 24-hour urine sodium | baseline to 12 months
  unadjusted and adjusted for creatinine excretion

SECONDARY OUTCOMES:
Change in 24-hour Ambulatory Systolic Blood Pressure | baseline to 12 months
Change in urine sodium/potassium ratio | baseline to 12 months
Change in Healthy Eating Index (HEI) score | baseline to 12 months
  Assessed by three 24-hour dietary recalls obtained by phone at each time point
Change in 24-hour Urine Albumin Excretion | baseline to 12 months
  unadjusted and adjusted for creatinine excretion
Change in weight | baseline to 12 months
Change in 24-hour urine phosphorus | baseline to 12 months
  unadjusted and adjusted for creatinine excretion
Change in Net Endogenous Acid Production (NEAP) | baseline to 12 months
  NEAP (mEq/d) = -10.2 + 54.5 (protein [g/d]/potassium [mEq/d])

CONTACTS AND LOCATIONS:
Overall Officials: Alex Chang, MD, Principal Investigator — Geisinger Clinic
Locations (2):
- United States (2):
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schrauben SJ, Inamdar A, Yule C, Kwiecien S, Krekel C, Collins C, Anderson C, Bailey-Davis L, Chang AR. Effects of Dietary App-Supported Tele-Counseling on Sodium Intake, Diet Quality, and Blood Pressure in Patients With Diabetes and Kidney Disease. J Ren Nutr. 2022 Jan;32(1):39-50. doi: 10.1053/j.jrn.2021.08.006. Epub 2021 Oct 11. PMID 34649784